CLINICAL TRIAL: NCT07384130
Title: Efficacy of Oral Probiotics on Cysteine-Induced Halitosis in Healthy Adult Volunteers.
Brief Title: Oral Probiotics for Halitosis in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John Hale (Industry)
Responsible Party: Sponsor-Investigator, John Hale, Chief Technology Officer, BLIS Technologies Limited
Organization: BLIS Technologies Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BLTCT2025/1; 2025EXP24497 (Other: Health and Disabilities Ethics Committee MOH Wellington NZ)
Record Dates: First submitted 2026-01-25; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Halitosis
Keywords: oral probiotic; halitosis; Streptococcus salivarius M18; Streptococcus salivarius K12; chewable tablet
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A staff member not part of the study group will be assigned to distribute blinded samples. The participant or the investigators will not be aware of the dose groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral probiotic lozenges (Active Comparator): Oral probiotic lozenges containing Streptococcus salivarius M18 and Streptococcus salivarius K12 and prebiotic
  Interventions: Dietary Supplement: In this study, a probiotic lozenge formulation containing S. salivarius K12, M18 and prebiotic will be evaluated for its potential to improve bad breath
- Placebo lozenges (Placebo Comparator): Oral lozenges
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: In this study, a probiotic lozenge formulation containing S. salivarius K12, M18 and prebiotic will be evaluated for its potential to improve bad breath — In this study, a probiotic-free lozenge formulation containing S. salivarius K12, M18 and prebiotic will be evaluated for its potential to improve bad breath as a comparator.
  Arms: Oral probiotic lozenges
Other: Placebo — Probiotic free placebo lozenge
  Arms: Placebo lozenges

SUMMARY:
The aim of this study is to evaluate efficacy of a probiotic lozenge containing BLIS M18, BLIS K12 and a prebiotic in healthy adults.

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled colonization pilot study with no crossover to evaluate the efficacy of probiotic lozenges on halitosis in healthy adults.

Participants will be randomly assigned to 2 groups consuming probiotic lozenge containing Streptococcus salivarius M18 and K12 and with prebiotic over a 13 day period. Breath scores will be measured at predetermined time points pre and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be otherwise healthy,
* practice good oral hygiene,
* 18 - 70 years of age

Exclusion Criteria:

* on antibiotic therapy,
* immunocompromised (have a weakened immune system)
* history of autoimmune disease,
* allergy or sensitivity to dairy,
* have an active periodontal disease, any known allergy or sensitivity to components of the test product or cysteine solution.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of Volatile Sulphur Compounds in ppb between the active and placebo groups | 13 days
  Study will determine the change in Volatile Sulphur Compounds (VSCs) as measured in ppb, following application of probiotic lozenges containing Streptococcus salivarius K12, Streptococcus salivarius M18 and prebiotic compared with a placebo lozenge. Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to post cysteine mouthrinse before the lozenge application and 13 days after once a day lozenge application with the level of significance of p≤0.05 across the probiotic and placebo lozenge. Appropriate statistical analysis software (e.g. Microsoft Excel) will be used to analyse the data

CONTACTS AND LOCATIONS:
Overall Officials: John R Tagg, PhD, Principal Investigator — BLIS Technologies Ltd
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data and information included in the Protocol and Clinical Study Report will be shared to other researchers and/or in publications in due course.
Supporting Information: Study Protocol, CSR
Time Frame: Study report 3 months after the completion of the study
Access Criteria: Summary study report will be shared by Principal Investigator upon request if not published in public literature

REFERENCES:
- [Background] Burton JP, Drummond BK, Chilcott CN, Tagg JR, Thomson WM, Hale JDF, Wescombe PA. Influence of the probiotic Streptococcus salivarius strain M18 on indices of dental health in children: a randomized double-blind, placebo-controlled trial. J Med Microbiol. 2013 Jun;62(Pt 6):875-884. doi: 10.1099/jmm.0.056663-0. Epub 2013 Feb 28. PMID 23449874